CLINICAL TRIAL: NCT02853695
Title: Implementation of Hysteroscopy in Flanders and the Netherlands
Status: Completed | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Dutch Society of Obstetricians and Gyneacologists (NVOG) (Unknown); Catharina Ziekenhuis Eindhoven (Other); Vlaamse Vereniging voor Obstetrie en Gynaecologie (Other)
Responsible Party: Sponsor
Organization: University Hospital, Ghent (Other)
Other Study IDs: B670201628466
Record Dates: First submitted 2016-07-19; First posted 2016-08-03 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Hysteroscopy; Minimally Invasive Surgical Procedures; Polyp; Myoma; Uterine Septum; Placental Remnant; Adhesiolysis
Keywords: Hysteroscopy; Diffusion; Implementation; Diagnostic hysteroscopy; Operative hysteroscopy
MeSH Terms: conditions — Polyps; Myoma; Septate Uterus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
By means of a questionnaire the investigators will study the implementation of hysteroscopy in Flanders and the Netherlands

DETAILED DESCRIPTION:
Hysteroscopy is a minimally invasive method for diagnosis and treatment of intra-uterine abnormalities. Complication and failure rates are low because of the direct visualisation of the treated abnormality. Moreover, hysteroscopic procedures replaced 'blind' (curettage) and more invasive interventions (hysterectomy).

The field of hysteroscopy has developed over the years. Changes occurred in hysteroscopic instruments and in the use of energy sources. An important development is the smaller diameter of the hysteroscopic system which makes it suitable for an outpatient setting. Not every gynaecologist, however, has the appropriate hysteroscopic skills or setting to carry out these procedures.

The incorporation of hysteroscopic procedures into daily practice in Flanders is unclear. In the Netherlands 2 surveys were conducted in the past to question the treatment options for polypectomy in an outpatient setting on the one hand and the diffusion of hysteroscopy on the other hand.

The investigators want to study the diffusion of hysteroscopy in Flanders and the Netherlands. Moreover the investigators want to provide an overview of the hysteroscopic procedures implemented, as well as the setting they are performed in.

An electronic questionnaire (LimeService) will be sent to all gynaecologists in Flanders and the Netherlands. Participation is voluntary and anonymous. After informed consent all gynaecologists are asked to complete the first part of the questionnaire containing general information. The second part is specific for gynaecologists performing hysteroscopy themselves, and inquires about the procedures they carry out.

ELIGIBILITY:
Inclusion Criteria:

* gynaecologist

Exclusion Criteria:

* residents in training for gynaecology/obstetrics

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Recognized gynaecologists (members of the Flemisch Society of Obstetricians and Gyneacologists (VVOG) and members of the Dutch Society of Obstetricians and Gyneacologists (NVOG))
Sampling Method: Non-Probability Sample
Enrollment: 249 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Questionnaire: Implementation of hysteroscopy | August 2016, questionnaire will be sent once at the start of the study
  the amount of gynaecologists performing hysteroscopy in relation to the total of gynaecologists participating in the questionnaire

SECONDARY OUTCOMES:
Questionnaire: setting for performing diagnostic hysteroscopy | August 2016, questionnaire will be sent once at the start of the study
  in which setting (office/operating room) diagnostic hysteroscopies are performed in relation to the total amount of diagnostic hysteroscopies performed
Questionnaire:Instrumentation used for hysteroscopy | August 2016, questionnaire will be sent once at the start of the study
  which instrumentation is used for specific hysteroscopic procedures.
Questionnaire: Diagnostic and techniques in the treatment of intrauterine pathology | August 2016, questionnaire will be sent once at the start of the study
  which diagnostics and techniques are used in the treatment of intrauterine pathology

CONTACTS AND LOCATIONS:
Overall Officials: Tjalina Hamerlynck, Study Director — Ghent University Hostpital

REFERENCES:
- [Background] Siristatidis C, Chrelias C, Salamalekis G, Kassanos D. Office hysteroscopy: current trends and potential applications: a critical review. Arch Gynecol Obstet. 2010 Oct;282(4):383-8. doi: 10.1007/s00404-010-1437-x. Epub 2010 Mar 27. PMID 20349076
- [Background] Valle RF. Development of hysteroscopy: from a dream to a reality, and its linkage to the present and future. J Minim Invasive Gynecol. 2007 Jul-Aug;14(4):407-18. doi: 10.1016/j.jmig.2007.03.002. PMID 17630157
- [Background] Timmermans A, van Dongen H, Mol BW, Veersema S, Jansen FW. Hysteroscopy and removal of endometrial polyps: a Dutch survey. Eur J Obstet Gynecol Reprod Biol. 2008 May;138(1):76-9. doi: 10.1016/j.ejogrb.2007.05.016. Epub 2007 Jul 12. PMID 17629392
- [Background] van Dongen H, Kolkman W, Jansen FW. Implementation of hysteroscopic surgery in The Netherlands. Eur J Obstet Gynecol Reprod Biol. 2007 Jun;132(2):232-6. doi: 10.1016/j.ejogrb.2006.04.016. Epub 2006 Jun 5. PMID 16737769
- [Background] Pascual-Pedreno A, Perez-Medina T, Brouard Urkiaga I, Fernandez-Parra J, Sobreviela-Laserrada M. Practice of endoscopic gynecologic surgery: a survey of Spanish gynecologists. Eur J Obstet Gynecol Reprod Biol. 2013 Jul;169(1):64-8. doi: 10.1016/j.ejogrb.2013.01.017. Epub 2013 Feb 21. PMID 23434402